CLINICAL TRIAL: NCT06792331
Title: Vaginal Natural Orifice Transluminal Surgery High Uterosacral Ligament Suspension Versus Laparoscopic Lateral Suspension in the Management of Vaginal Vault Prolapse: Initial Experience in a Single Center With a Median-term Follow-up
Brief Title: Vaginal Vault Prolapse Surgical Treatment
Acronym: VVPST
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arzu Bilge Tekin, Assoc. Prof. MD, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: VVPST
Record Dates: First submitted 2025-01-11; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Vaginal Vault Prolapse; Pelvic Floor Prolapse
Keywords: Vaginal vault prolapse; vNOTES; high uterosacral ligament suspension; lateral suspension; laparoscopy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women with vNOTES high uterosacral ligament suspension: Symptomatic women aged 40-80 years old with ≥ stage 2 vault prolapse who underwent vNOTES high uterosacral ligament suspension and laparoscopic lateral suspension.
  Interventions: Procedure: vNOTES high uterosacral ligament suspension
- Women with laparoscopic lateral suspension.: Symptomatic women aged 40-80 years old with ≥ stage 2 vault prolapse who underwent laparoscopic lateral suspension.
  Interventions: Procedure: Laparoscopic lateral suspension

INTERVENTIONS:
Procedure: vNOTES high uterosacral ligament suspension — Following the entry into the peritoneal cavity via apical colpotomy, a transvaginal retractor was inserted through the vaginal vault and the vaginal access platform was established. The ureters and uterosacral ligaments (USL) were identified via laparoscopic view. Bilateral nonabsorbable sutures were placed by the intermediate portions of the USL at the level of the ischial spines making up a total of 4 stitches (Figure 1). Then, the sutures were slightly weighed to verify proper placement. Then, the V-notes platform was removed and the peritoneum was closed. The aforementioned sutures were fixed to the ipsilateral cardinal ligament stump and the pubocervical fascia on the anterior wall. Finally, the previously mentioned nonabsorbable sutures were attached to the vaginal cuff and tied. Routine postoperative cystoscopy was performed.
  Groups: Women with vNOTES high uterosacral ligament suspension
Procedure: Laparoscopic lateral suspension — The polypropylene mesh used had a width of 2.5 cm and a length of 25 cm. The vaginal cuff was suspended. Blunt dissection was applied to develop vesicovaginal and rectovaginal spaces. The middle part of the mesh was placed flatly in the vesicovaginal space, and fixed with non-absorbable sutures. An atraumatic laparoscopic instrument was inserted through skin incisions of approximately 2-3 mm approximately 3 cm above and 4 cm lateral to the anterior superior iliac spine, followed by perforation only of the aponeurosis of the external oblique muscle and retroperitoneal advancement of the instrument through the lateral abdominal wall. Under laparoscopic visualization, the instrument moved through the bilateral tension-free retroperitoneal tunnels created. The lateral arms of the mesh were secured bilaterally to the aponeurosis of the external oblique muscle and behind the anterior superior iliac spine. Finally, the peritoneum was closed.
  Groups: Women with laparoscopic lateral suspension.

SUMMARY:
Since apical support is the mainstay of vaginal cuff restoration, sacrocolpopexy is still accepted as the gold standard technique in vaginal vault prolapse (VVP). The increased risk of surgical morbidity in the abdominal approach has prompted the interest in minimally invasive surgery. Laparoscopic lateral suspension (LLS) using mesh is an efficient alternative technique for apical support. In addition, vaginal approaches have been used in cuff prolapsus surgery for many years. Uterosacral ligaments are strong native tissues used in cuff surgery and apical support. In recent years, Vaginal Natural Orifice Transluminal Endoscopic Surgery (VNOTES) has offered advantages particularly complications related to the ureter over the traditional transvaginal uterosacral ligament suspension in cuff restoration.

DETAILED DESCRIPTION:
Hysterectomy is one of the common surgical procedures in current gynecology practice and is a risk factor for vault prolapse. Since apical support is the mainstay of vaginal cuff restoration, sacrocolpopexy is still accepted as the gold standard technique in vaginal vault prolapse (VVP). The increased risk of surgical morbidity in the abdominal approach has prompted the interest in minimally invasive surgery. Laparoscopic lateral suspension (LLS) using mesh is an efficient alternative technique for apical support. In addition, vaginal approaches have been used in cuff prolapsus surgery for many years. Uterosacral ligaments are strong native tissues used in cuff surgery and apical support. In recent years, Vaginal Natural Orifice Transluminal Endoscopic Surgery (VNOTES) has offered advantages particularly complications related to the ureter over the traditional transvaginal uterosacral ligament suspension in cuff restoration. Lack of incision pain, better cosmetic results, and direct visualization of important structures such as the rectum and ureter that cannot be obtained with the traditional transvaginal approach are important advantages of vNOTES approach.

ELIGIBILITY:
Inclusion Criteria:

* Women with vaginal vault prolapse

Exclusion Criteria:

* Women who have previously undergone surgical treatment for pelvic organ prolapse
* Women who needed additional surgery due to anterior or posterior prolapse or stress incontinence
* Pelvic inflammatory disease
* Suspected gynecological malignancy
* Rectovaginal endometriosis
* obliterated rectovaginal space detected on pelvic examination.

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with vaginal vault prolapse
Study Population: Symptomatic women aged 40-80 years old with ≥ stage 2 vault prolapse who underwent vNOTES high uterosacral ligament suspension and laparoscopic lateral suspension
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Anatomical and functional outcomes | 14-30 months
  Evaluation of Pelvic organ prolapse quantification (POP-Q) scores before and after surgeries.
  Clinical assessment of the pelvic floor was performed by a gynecologist experienced in the evaluation of pelvic organ prolapse, while patients were in the supine lithotomy position. In the POP-Q, nine measurement points are assessed during the maximal Valsalva maneuver, except for the transvaginal length (TVL), measured at rest. Only the measurements of POP-Q points Ba, C, Bp were used to compare preoperative and postoperative evaluation. Ba is the most descended edge on the anterior vaginal wall, C represents either the most distal edge of the cervix or the leading edge of the vaginal vault, Bp is the most descended edge on the posterior vagina wall. Measurements in centimeters relative to the hymenal remnants were used in the analysis.
Requirement of reoperation | 14-30 months
  Number and rate of women requiring subsequent surgery for pelvic organ prolapse following the studied surgeries.
Subjective recurrence | 14-30 months
  The presence of bulging symptoms

SECONDARY OUTCOMES:
Transition of patient condition after surgery | 6 months
  Patient Global Impression of Improvement (PGI-I) is a transition scale that is a single question asking the patient to rate their pelvic organ prolapsus condition now, as compared with how it was before beginning treatment on a scale from 1. Very much better to 7. Very much worse.
Sexual Function | 6 months
  Validated versions of Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and Female Sexual Function Index (FSFI) questionnaire11,12 are routinely applied preoperatively and at 6 months postoperatively
Change in quality of life | 6 months
  A seven-point quality of life (QoL) questionnaire ranging from 1 (very much improved) to 7 (very much worse), was used to assess patients' postoperative satisfaction
Change of sexual function | 6 months
  Female Sexual Function Index (FSFI) questionnaire are routinely applied preoperatively and at 6 months postoperatively. The FSFI is a survey measuring the sexual functioning of women in six different domains: desire, arousal, lubrication, orgasm, satisfaction and pain. Each item is scored from 0 to 5 except for questions 1, 2, 13-16 (which are scored from 1 to 5).
  The 19 items of the FSFI use a 5-point Likert scale ranging from 1-5 with higher scores indicating greater levels of sexual functioning on the respective item. To score the measure, the sum of each domain score is first multiplied by a domain factor ratio (0.6 for desire; 0.3 for arousal; 0.3 for lubrication; 0.4 for orgasm; 0.4 for satisfaction; and 0.4 for pain) to place all domains totals on a more comparable scale, and then subsequently summed to derive a total FSFI score.
Parameters regarding surgery | 14-30 months
  Duration of surgery in minutes,preoperative-postoperative hemoglobin difference (g/dL), postoperative length of hospital stay (day), number of hospital readmissions after discharge from hospital, intraoperative and postoperative complications via Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu B Tekin, Study Chair — SBÜ Sancaktepe Şehit Prof Dr İlhan Varank EAH
Locations (1):
- Arzu Bilge Tekin, Istanbul, Sancaktepe, Turkey (Türkiye)

REFERENCES:
- [Background] Lu Z, Chen Y, Wang X, Li J, Hua K, Hu C. Transvaginal natural orifice transluminal endoscopic surgery for uterosacral ligament suspension: pilot study of 35 cases of severe pelvic organ prolapse. BMC Surg. 2021 Jun 8;21(1):286. doi: 10.1186/s12893-021-01280-6. PMID 34103032
- [Background] Lowenstein L, Baekelandt J, Paz Y, Lauterbach R, Matanes E. Transvaginal Natural Orifice Transluminal Endoscopic Hysterectomy and Apical Suspension of the Vaginal Cuff to the Uterosacral Ligament. J Minim Invasive Gynecol. 2019 Sep-Oct;26(6):1015. doi: 10.1016/j.jmig.2019.04.007. Epub 2019 Apr 10. PMID 30980991
- [Background] Dubuisson J, Veit-Rubin N, Bouquet de Joliniere J, Dubuisson JB. Laparoscopic Lateral Suspension: Benefits of a Cross-shaped Mesh to Treat Difficult Vaginal Vault Prolapse. J Minim Invasive Gynecol. 2016 Jul-Aug;23(5):672. doi: 10.1016/j.jmig.2016.01.028. Epub 2016 Feb 8. PMID 26867700